CLINICAL TRIAL: NCT02123277
Title: Long Term Evaluation of Tubal Expansion on Obstructive Dysfunctions of Eustachian Tube
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9259
Record Dates: First submitted 2014-03-03; First posted 2014-04-25 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Eustachian Tube Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- concept proof (Experimental): Balloon catheter for the Eustachian tube
  Interventions: Device: Balloon catheter for the Eustachian tube

INTERVENTIONS:
Device: Balloon catheter for the Eustachian tube — Balloon catheter is inserted in the Eustachian tube to dilate it.

SUMMARY:
The study aim is to evaluate the tubal score on patients who suffer from obstructive dysfunction of eustachian tube before and after the eustachian tube dilatation.

DETAILED DESCRIPTION:
The study aim is to evaluate the tubal score on patients who suffer from obstructive dysfunction of eustachian tube before the intervention and 12 months after the eustachian tube dilatation.

This patients are refractory to the reference medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients between 20 and 80 years old
* tubal score lower than 5
* patients who already used reference medical treatment

Exclusion Criteria:

* patients who already do a major surgery of middle ear
* tympanic perforation
* pregnant or breastfeeding woman.
* patients who can't be follow during 14 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-05; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in Tubal score | at 1st day, and 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Frederic VENAIL, Principal Investigator — CHRU Montpellier
Locations (1):
- Gui de Chauliac Hospital, Montpellier, France

REFERENCES:
- [Derived] Swords C, Smith ME, Patel A, Norman G, Llewellyn A, Tysome JR. Balloon dilatation of the Eustachian tube for obstructive Eustachian tube dysfunction in adults. Cochrane Database Syst Rev. 2025 Feb 26;2(2):CD013429. doi: 10.1002/14651858.CD013429.pub2. PMID 40008607
- [Derived] Kaderbay A, Karkas A, Schmitt D, Mura T, Lavieille JP, Venail F. Balloon dilation for persistent unilateral chronic obstructive Eustachian tube dysfunction is effective: a prospective multicentre study. Eur Arch Otorhinolaryngol. 2023 Mar;280(3):1101-1109. doi: 10.1007/s00405-022-07578-2. Epub 2022 Aug 6. PMID 35932313